CLINICAL TRIAL: NCT01343901
Title: A Cohort Study of Patients With Metastatic Colorectal Cancer Treated With Avastin® as First-line Therapy for Liver Metastases Considered as Potentially Resectable
Brief Title: An Observational Study on Bevacizumab (Avastin) as First-Line Treatment in Colorectal Cancer Participants With Potentially Resectable Liver Metastases
Acronym: PICASSO
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22999
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Bevacizumab: Participants with metastatic colorectal cancer (mCRC) with exclusively liver or liver and lung metastases, who were receiving bevacizumab as part of first line treatment for potentially resectable liver metastases will be observed.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Participants with mCRC and having exclusively liver or liver and lung metastases who were receiving bevacizumab as part of first line treatment for potentially resectable liver metastases as per treating physician's discretion will be observed. All concomitant medications as used in routine clinical practice are allowed.
  Other Names: Avastin

SUMMARY:
This observational study will evaluate the efficacy and safety of bevacizumab as first-line treatment in participants with colorectal cancer and potentially resectable liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Participants with colorectal cancer with exclusively hepatic or hepatic and pulmonary metastases
* First-line treatment with bevacizumab for potentially resectable metastatic disease

Exclusion Criteria:

* Outright resectable disease
* Clearly inoperable disease
* Participation in a clinical trial evaluating a cytotoxic anticancer treatment and/or an innovative therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with colorectal cancer and hepatic or hepatic and pulmonary metastases
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (126):
- France (126):
  - Clinique Esquirol Saint Hilaire, Agen
  - C.H. Du Pays D'aix En Provence Service du Dr Blanc, Aix-en-Provence
  - Poly Parc Rambot La Provencale; Chimiotherapie Ambulatoire, Aix-en-Provence
  - Chi D Alencon; Medecine Ambulatoire, Alençon
  - Ch D Ales; Oncologie, Alès
  - Hopital Nord; Medecine A, Amiens
  - Clinique De L Europe; Pmsi, Amiens
  - Clinique De L Europe; Radiotherapie Chimiotherapie, Amiens
  - Centre Hospitalier de L'Agglomeration Montargeoise; Medecine Polyvalente A Orientation Mi & Cancero, Amilly
  - Hotel Dieu; Medecine A, Angers
  - Centre Radiotherapie Marie Curie, Arras
  - HOP Prive Arras Les Bonnettes; Chimiotherapie, Arras
  - Polyclinique Sainte Marguerite; Chimiotherapie, Auxerre
  - Chic Cote Basque Bayonne; Medecine II, Bayonne
  - Clinique Saint Etienne; Medecine, Bayonne
  - Centre Hospitalier; Hematologie-Oncologie, Beauvais
  - Ch de Belfort; Hopital de Jour, Belfort
  - Hopital Jean Minjoz; Gastro Enterologie, Besançon
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Centre Pierre Curie, Beuvry
  - Centre De Radiotherapie Oncodoc, Béziers
  - Clinique Champeau Mediterranee; Radiotherapie Oncologie, Béziers
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Fondation Bergonie; Gastro-Enterologie, Bordeaux
  - Polyclin Bordeaux Nord Aquitaine; Gastro Enterologie, Bordeaux
  - Clinique Du Docteur Convert; Medecine, Bourg-en-Bresse
  - Centre Hospitalier Fleyriat; Oncologie/Hematologie, Bourg-en-Bresse
  - Ch De Fleyriat; Gastro Enterologie, Bourg-en-Bresse
  - Ch Pierre Oudot; Gastro Enterologie, Bourgoin
  - Ch Jean Rougier; Oncologie Gastro Enterologie, Cahors
  - Infirmerie Protestante; Endos Digestive Coelioscopie, Caluire-et-Cuire
  - Ch Antoine Gayraud; Oncologie, Carcassonne
  - Cabinet Medical, Challes-les-Eaux
  - Ch de Chambery; Gastro Enterologie, Chambéry
  - Hopital Manchester; Gastro Enterologie, Charleville-Mézières
  - CH Du Cotentin Site De Cherbourg; Hopital De Jour, Cherbourg Octeville
  - Clinique Des Cedres; Medecine 2, Cornebarrieu
  - CHU Henri Mondor; Service d'Oncologie Medicale, Créteil
  - Ch De Dax; Radiotherapie Oncologie, Dax
  - Centre Leonard De Vinci;Chimiotherapie, Dechy
  - Cabinet, Dijon
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Ch De La Dracenie; Hopital De Jour, Draguignan
  - Hopital Victor Jousselin; Gastro Enterologie, Druex
  - Hopital Simone Veil Eaubonne; Hopital De Jour, Eaubonne
  - Clinique Pasteur; Oncologie Medicale, Hematologie, Évreux
  - Ch Jacques Monod;Medecine A4 B4, Flers
  - Hopital De Freyming; Secteur 1, Freyming-Merlebach
  - Centre Gastro Loire, Gien
  - Hopital Nord Ouest;Gastro Enterologie, Gleizé
  - Hopital Alpha Sante De Hayange; Medecine B, Hayange
  - Clinique de L' Esperance; Oncologie, Hyères
  - Clinique Sainte Marguerite; Oncologie Medicale, Hyères
  - Polyclinique de Blois; Chimiotherapie Ambulatoire, La Chaussée-Saint-Victor
  - CH Dptal Les Oudairies; Gastro Enterologie, La Roche-sur-Yon
  - CH Dptal Les Oudairies; Hematologie Oncologie, La Roche-sur-Yon
  - Hopital Albert Michallon; Gastro Enterologie, La Tronche
  - Hopital Albert Michallon; Radiotherapie, La Tronche
  - Hopital Robert Boulin; Oncologie, Libourne
  - Cabinet Medical, Lille
  - Clinique Chenieux; Oncology, Limoges
  - Ch De Longjumeau; Hopital De Jour Et Semaine, Longjumeau
  - CH Bretagne Sud Site Bodelio; Oncologie Radiotherapie, Lorient
  - Clinique Des 4 Pavillons; Chimiotherapie, Lormont
  - Hia Desgenettes; Oncologie Hematologie, Lyon
  - Hopital De La Croix Rousse;Hepato Gastro Entero, Lyon
  - Clinique De La Sauvegarde; Chimiotherapie, Lyon
  - Ctre Hosp St Joseph Et St Luc; Gastro Enterologie Endoscopie, Lyon
  - Hopital Prive Jean Mermoz; Cancerologie, Lyon
  - Clinique Saint Faron; Sce Oncologie Radiotherapie, Mareuil-lès-Meaux
  - Fondation Hopital Saint Joseph; Gastro-Enterologie, Marseille
  - Ch De Meaux; Gastro Enterologie, Meaux
  - Hopital Clinique Claude Bernard; Oncologie Medicale, Metz
  - Chra; Gastro Enterologie, Metz-Tessy
  - Hopital Layne; Medecine Ambulatoire, Mont-de-Marsan
  - Site Le Mittan; Hopital De Jour, Montbéliard
  - Ch De Montelimar; Gastro Enterologie Oncologie, Montélimar
  - Ghi Le Raincy Montfermeil; Gastro Medecine Interne, Montfermeil
  - Ghi Le Raincy Montfermeil; Radiotherapie Oncologie, Montfermeil
  - Ctre Radiotherapie Joseph Belot; Hematologie, Montluçon
  - Polyclinique Saint Roch; Hop Jour Chimio Radiotherapie, Montpellier
  - Centre Azureen De Cancerologie; Cons externes, Mougins
  - Polyclinique Gentilly; CHIMIOTHERAPIE AMBULATOIRE, Nancy
  - Polyclinique Du Languedoc; Chimiotherapie, Narbonne
  - Ch De Nemours; Medecine 1, Nemours
  - Clinique Du Parc Imperial; Chimiotherapie, Nice
  - Hopital De L Archet;Gastro Nutrition Oncologie, Nice
  - Hopital Caremeau; Gastro Enterologie, Nîmes
  - Hopital Des Diaconesses; Hopital De Jour, Paris
  - Ch Pitie Salpetriere; Oncologie Medicale, Paris
  - GH Paris Saint Joseph; Hopital De Jour Oncologie, Paris
  - Hopital Bichat Claude Bernard; Hepatologie Gastro Enterologie, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Centre Catalan D' Oncologie, Perpignan
  - Hopital Saint Jean; Centre Henri Pujol, Perpignan
  - Hopital Du Haut-Leveque; Gastro-Enterologie, Pessac
  - Clinique Francheville; Radiotherapie, Périgueux
  - Ch De Perigueux; Had Perigueux, Périgueux
  - Ch Lyon Sud; Gastro Secteur Jules Courmont, Pierre-Bénite
  - Clinique Armoricaine Radiologie; Hopital de Jour, Plérin
  - Chu La Miletrie; Gastro Enterologie Endoscopies, Poitiers
  - Hopital Rene Dubos; Service de Medecine Generale & de Gastro-Enterologie, Pontoise
  - Centre Eugene Marquis; Unite Huguenin, Rennes
  - Hopital Charles Nicolle; Endoscopies Digestives, Rouen
  - Clinique De L Europe; Chimiotherapie, Rouen
  - Clinique Saint Hilaire; Sce Chimiotherapie, Rouen
  - Hopital Yves Le Foll; Hepatologie Gastro Enterologie, Saint-Brieuc
  - Chi Poissy Saint Germain En Laye; Centre Coordination Cancerologie, Saint-Germain-en-Laye
  - Chp Saint Gregoire; Cancerologie Radiotherapie, Saint-Grégoire
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Clinique de L'Union; Oncologie, Saint-Jean
  - Memorial France Etats Unis; Hopital De Jour, Saint-Lô
  - CMCO De La Cote D Opale; Auberge De Jour, Saint-Martin-Boulogne
  - Cabinet Medical, Saint-Priest
  - Centre Hospitalier General; Oncologie Medicale, Salouël
  - Clinique Chir De L Orangerie; Chimiotherapie, Strasbourg
  - Clinique Saint Anne; Hopital De Jour, Strasbourg
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Clinique Sainte Anne; Hospitalisation, Strasbourg
  - Hopital Font Pre; Hemato-Oncologie, Toulon
  - Hopital Purpan; Chir Generale Digestive, Toulouse
  - Clinique Pasteur; Oncologie Medicale, Toulouse
  - Hopital Saint Nicolas; Medecine A, Verdun
  - Hopital Jacques Lacarin; Hopital De Jour, Vichy
  - Hopital Paul Brousse; Hematologie, Villejuif
  - Chi De Villeneuve St Georges; Oncologie, Villeneuve-Saint-Georges

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: All participants with metastatic colorectal cancer (mCRC) with exclusively liver or liver and lung metastases for whom bevacizumab (Avastin) was administered as part of first line treatment for potentially resectable liver metastases as per treating physician discretion. All concomitant medications as used in daily routine clinical practice were allowed.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 210
Efficacy Population | 205
Completed | 97
Not Completed | 113
Not completed — Death | 85
Not completed — Physician Decision | 4
Not completed — Lost to Follow-up | 12
Not completed — Management by another medical team | 11
Not completed — Participant decision | 1

BASELINE CHARACTERISTICS:
Population: Efficacy population included all participants having at least one dose of bevacizumab without protocol deviations.
Groups:
- Bevacizumab: All participants with mCRC with exclusively liver or liver and lung metastases, who were receiving bevacizumab as part of first line treatment for potentially resectable liver metastases as per treating physician's discretion were observed. All concomitant medications as used in routine clinical practice were allowed.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.83 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 132

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Detectable Metastatic Disease After Secondary Resection Post Surgery
Description: Secondary resection involves removal of all detectable metastases at surgery including participants with missing metastases left in place. Percentage of participants without detectable metastatic disease after secondary resection removing all detectable metastases at surgery (including participants with disappeared metastases left in place [missing metastases]) was reported. Metastases was detected using computed tomography (CT) scan or magnetic resonance imaging (MRI).
Time Frame: Baseline up to 36 months
Population: Efficacy population. Here number of participants analyzed represents the number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 104
Percentage of participants | 84.6

2. Primary Outcome: Percentage of Participants Without Detectable Metastatic Disease After a Complete Response Without Surgery
Description: The percentage of participants with no detectable metastatic disease after a complete response without surgery (missing metastasis) was reported.
Time Frame: Baseline up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 90
Percentage of participants | 4.4

3. Secondary Outcome: Percentage of Participants With at Least One Disease and Comorbidity at Day 0
Description: Percentage of participants who had any concurrent disease (comorbidity) at Day 0 was reported. Comorbidities included gastrointestinal disease, hypertension, other cardiovascular disease, and other medical history and comorbidities (other than those specified above). Same participant may be counted in more than one category.
Time Frame: Day 0
Population: Efficacy population. Here number of participants analyzed represents the number of participants evaluable for this outcome and 'n' represents the number of participants available for assessment at a given category.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 204
Percentage of participants
  Gastrointestinal disease (n=201) | 7.5
  Hypertension (n=202) | 41.6
  Other cardiovascular disease (n=202) | 13.9
  Other medical history and comorbidities (n=204) | 52.9

4. Secondary Outcome: Percentage of Participants With Different Previous Therapies at Day 0
Description: Previous therapies included neoadjuvant treatment (chemotherapy or chemotherapy + radiotherapy) and adjuvant treatment (FOLFOX [folinic acid+5-fluorouracil+oxaliplatin], LV5FU2 [leucovorin+5-Fluorouracil], capecitabine, or any other adjuvant treatment). Only participants who received neoadjuvant treatment and adjuvant treatment was reported.
Time Frame: Day 0
Population: Efficacy population. Here number of participants analysed represents the number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 55
Percentage of participants
  With Neoadjuvant Treatment | 29.1
  With Adjuvant Treatment | 52.7

5. Secondary Outcome: Mean Number of Cumulated Cycles of Bevacizumab Over the Study Period
Time Frame: Baseline up to 36 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cycles
Arm/Group | Bevacizumab
Number analyzed (Participants) | 191
Cycles | 14.40 (10.80)

6. Secondary Outcome: Percentage of Participants Who Received at Least One Chemotherapy Over the Study Period
Time Frame: Baseline up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 181
Percentage of participants | 96.1

7. Secondary Outcome: Percentage of Participants With at Least One Comorbidity Post Bevacizumab Treatment
Description: Percentage of participants who had any concurrent disease (comorbidity) was reported. Comorbidities included gastrointestinal disease, other cardiovascular disease, and other medical history and comorbidities (other than those which are specified above). Same participant may be counted in more than one category.
Time Frame: Baseline up to 36 months
Population: Analysis population consisted of participants with disappeared metastasis left in place with or without surgery. Here number of participants analyzed represents the number of participants evaluable for this outcome and 'n' represents the number of participants available for assessment at a given category.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 92
Percentage of participants
  Gastrointestinal disease | 8.0
  Other cardiovascular disease | 10.9
  Other medical history and comorbidities | 54.9
  Respiratory, thoracic and mediastinum disorders | 4.0

8. Secondary Outcome: Percentage of Participants With Disease Progression or Death
Description: Disease progression is defined at least a 20 percent (%) increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 millimeter (mm) or persistence of non-target lesions, or appearance of one or more new lesions.
Time Frame: Baseline until disease progression or death, whichever occurred first, assessed up to 36 months
Population: Efficacy population
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 205
Percentage of participants | 82.9

9. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival defined as the time elapsed between the Avastin start date and the date of first progressive disease (PD) or death. Kaplan-Meier estimate was used for evaluation. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions or appearance of one or more new lesions.
Time Frame: Baseline until disease progression or death, whichever occurred first, assessed up to 36 months
Population: Efficacy population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 205
Months | 11.50 [10.38 to 12.35]

10. Secondary Outcome: Percentage of Participants With Disease Relapse
Description: Relapse was defined as the presence of metastases post last surgery removing all detectable metastases (A1 criterion [participants without detectable metastatic disease {DMD} after secondary resection removing all detectable metastases at surgery {including participants with missing metastases}]) and the date of first PD or death. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions, or appearance of one or more new lesions.
Time Frame: Baseline until disease progression or death, whichever occurred first, assessed up to 36 months
Population: Efficacy population. Here number of participants analyzed signifies efficacy population with surgery removing all the detectable metastases.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 88
Percentage of participants | 76.1

11. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS was defined as the time elapsed between the last surgery removing all detectable metastases (A1 criterion [participants without DMD after secondary resection removing all detectable metastases at surgery {including participants with missing metastases}]) and the date of first PD or death. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions, or appearance of one or more new lesions.
Time Frame: Baseline until disease progression or death, whichever occurred first, assessed up to 36 months
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 88
Months | 11.10 [7.82 to 14.62]

12. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Baseline until death; assessed up to 36 months
Population: Efficacy population
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 205
Percentage of participants | 41.0

13. Secondary Outcome: Overall Survival (OS)
Description: OS time is defined as time between start of therapy and date of death. Kaplan-Meier estimate was used for evaluation.
Time Frame: Baseline until death, assessed up to 36 months
Population: Efficacy population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 205
months | NA [NA to NA] — Survival time was not reached due to high number of censored participants.

14. Secondary Outcome: Percentage of Participants With Histologically Viable Tumor Cells With Resected Non Detectable Hepatic and Pulmonary Metastases Post Surgery
Description: For the non-detectable liver and lung metastases the categorization based on rate of viable cells were as follows (no viable cells =0%, minimum =1 to 49%, maximum =50 to 100%).
Time Frame: Baseline up to 36 months
Population: Efficacy population. Here number of participants analyzed represents the overall number of participants evaluable for this outcome and 'n' represents the number of participants available for assessment at a given category.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 104
Percentage of participants
  Hepatic metastases:No viable cell (0%)(n=70) | 4.3
  Hepatic metastases:Minimum (1 - 49 %)(n=70) | 8.6
  Hepatic metastases:Maximum (>=50%)(n=70) | 7.1
  Hepatic metastases:Not Applicable(n=70) | 80.0
  Pulmonary metastases:Maximum (>=50%)(n=80) | 1.3
  Pulmonary metastases:Not Applicable(n=80) | 98.8

15. Secondary Outcome: Number of Cumulated Cycles of First Line Bevacizumab at Day 0
Time Frame: Day 0
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Bevacizumab
Number analyzed (Participants) | 195
cycles | 10.20 (7.79)

16. Secondary Outcome: Percentage of Participants With Different Doses of First Line Bevacizumab at Day 0
Time Frame: Day 0
Population: Efficacy population. Here, number of participants analyzed represents the number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 196
Percentage of participants
  5 milligrams per kilogram (mg/kg)/2 weeks | 94.9
  7.5 mg/kg/3 weeks | 3.1
  10 mg/kg/2 weeks | 2.0

17. Secondary Outcome: Total Duration of First Line Bevacizumab Treatment at Day 0
Time Frame: Day 0
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 195
months | 4.67 [0.5 to 33.2]

18. Secondary Outcome: Percentage of Participants With Unresectability Criteria
Time Frame: Day 0
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 201
Percentage of participants
  Oncological Reason (n=201) | 81.6
  Technical Reason (n=191) | 12.0
  Both Oncological and Technical Reason (n=191) | 10.5

ADVERSE EVENTS:
Time Frame: Baseline up to 36 months
Description: Safety population included all participants with at least one dose of bevacizumab.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 71/210
Other Adverse Events (participants affected / at risk) | 75/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=210)
Diarrhoea (Gastrointestinal disorders) | 4
Subileus (Gastrointestinal disorders) | 3
Gastrointestinal obstruction (Gastrointestinal disorders) | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Colonic fistula (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Infectious peritonitis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 4
Sepsis (Infections and infestations) | 3
Device related infection (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Sepsis syndrome (Infections and infestations) | 1
General physical health deterioration (General disorders) | 6
Chills (General disorders) | 1
Death (General disorders) | 1
Hyperthermia (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Aortic thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Transient ischaemic attack (Vascular disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Vascular injury (Injury, poisoning and procedural complications) | 1
Renal failure (Renal and urinary disorders) | 2
Bladder dilatation (Renal and urinary disorders) | 1
Bladder obstruction (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Biliary fistula (Hepatobiliary disorders) | 1
Biloma (Hepatobiliary disorders) | 1
Chronic hepatic failure (Hepatobiliary disorders) | 1
Hepatic atrophy (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Aphasia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Completed suicide (Psychiatric disorders) | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=210)
Asthenia (General disorders) | 44
Mucosal inflammation (General disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 37
Nausea (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 12
Paraesthesia (Nervous system disorders) | 20
Neuropathy peripheral (Nervous system disorders) | 16
Neutropenia (Blood and lymphatic system disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 12
Hypertension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.